CLINICAL TRIAL: NCT02537574
Title: A Phase 3 Study to Evaluate the Safety, Tolerability, and Efficacy of Naltrexone for Use in Conjunction With Buprenorphine in Adults With Opioid Use Disorder Prior to First Dose of VIVITROL®
Brief Title: Naltrexone for Use in Conjunction With Buprenorphine in Adults With Opioid Use Disorder Prior to First Dose of VIVITROL® (Naltrexone for Extended-Release Injectable Suspension)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALK6428-A301
Record Dates: First submitted 2015-08-31; First posted 2015-09-01 (Estimated); Results first posted 2019-01-09 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Opioid Use Disorder
Keywords: Alkermes; Buprenorphine; Naltrexone; Vivitrol; Opioid Use; Opiates; Dependence; Abuse; Heroin; Painkillers; Substance Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NTX/BUP (Experimental): Oral naltrexone + sublingual buprenorphine
  Interventions: Drug: NTX/BUP
- NTX/PBO-B (Active Comparator): Oral naltrexone + sublingual placebo
  Interventions: Drug: NTX/PBO-B
- PBO-N/PBO-B (Placebo Comparator): Oral placebo naltrexone + sublingual placebo buprenorphine
  Interventions: Drug: PBO-N/PBO-B

INTERVENTIONS:
Drug: NTX/BUP — Daily doses
  Arms: NTX/BUP
Drug: NTX/PBO-B — Daily doses
  Arms: NTX/PBO-B
Drug: PBO-N/PBO-B — Daily doses
  Arms: PBO-N/PBO-B

SUMMARY:
This study will evaluate the safety, effectiveness and tolerance of low doses of oral naltrexone along with buprenorphine to treat opioid use disorder prior to the first injection of VIVITROL.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Willing and able to provide government-issued identification
* Has a BMI of 18.0-40.0 kg/m^2
* Has a physiologic dependence on opioids
* Is voluntarily seeking treatment for opioid use disorder and willing to completely withdraw from his/her opioid use throughout the study with desire for or motivation for antagonist therapy
* Wiling to abide by the contraception requirements for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Is pregnant, planning to become pregnant or breastfeeding during the study
* Has used Buprenorphine within 7 days prior to randomization
* Has used Methadone within 14 days prior to randomization
* Has a history of VIVITROL use within 90 days prior to screening or has used oral naltrexone within 14 days prior to randomization
* Has a history of seizures or has received anticonvulsant therapy within the past 5 years
* Has a condition, disease state, or previous medical history that would preclude safe participation in the study or affect the ability to adhere to the protocol visit schedule, requirements, or assessments
* Has a current diagnosis of schizoaffective disorder, bipolar disorder, or untreated and unstable major depressive disorder
* Is currently physiologically dependent on any psychoactive substance (except opioids, caffeine, or nicotine) requiring medical intervention for detoxification
* Has a history of hypersensitivity or adverse reaction to Buprenorphine, Naltrexone, or Naloxone
* Has a history of more than 3 unsuccessful inpatient or medically assisted outpatient opioid detoxifications during his/her lifetime
* Has significant suicidal ideation or behavior within the past year
* Is currently participating, or has participated, in a clinical trial of an investigational drug, device, or biologics within 3 months prior to screening
* Has a history of accidental opioid drug overdose in the past 3 years whether or not medical treatment was sought or received
* Is court mandated to receive treatment for opioid use disorder
* Additional criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2017-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Sullivan, MD, PhD, Study Director — Alkermes, Inc.
Locations (20):
- United States (20):
  - North Country Clinical Research, Oceanside, California
  - NRC Research Institute, Orange, California
  - Atlantic Shores Hospital, Lauderhill, Florida
  - TRY Research, Maitland, Florida
  - Research Centers of America, Oakland Park, Florida
  - CNS Healthcare, Orlando, Florida
  - Neuroscience Research Institute, Winfield, Illinois
  - John Hopkins University School of Medicine, Baltimore, Maryland
  - Comprehensive Clinical Research, Berlin, New Jersey
  - PRA Health Sciences, Marlton, New Jersey
  - New York State Psychiatric Institute/ Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - University Of Pennsylvania - Treatment Research Center, Philadelphia, Pennsylvania
  - Western Psychiatric Institute and Clinic of UPMC, Pittsburgh, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas
  - Insite Clinical Research, DeSoto, Texas
  - Baylor College of Medicine, Houston, Texas
  - Pharmaceutical Research Associates Inc., Salt Lake City, Utah

REFERENCES:
- [Result] Bisaga A, Mannelli P, Yu M, Nangia N, Graham CE, Tompkins DA, Kosten TR, Akerman SC, Silverman BL, Sullivan MA. Outpatient transition to extended-release injectable naltrexone for patients with opioid use disorder: A phase 3 randomized trial. Drug Alcohol Depend. 2018 Jun 1;187:171-178. doi: 10.1016/j.drugalcdep.2018.02.023. Epub 2018 Apr 10. PMID 29674251
- [Derived] Mannelli P, Douaihy AB, Zavod A, Legedza A, Akerman SC, Sullivan MA. Patterns of withdrawal in patients with opioid use disorder (OUD) transitioning from untreated OUD or buprenorphine treatment to extended-release naltrexone. Am J Drug Alcohol Abuse. 2021 Nov 2;47(6):753-759. doi: 10.1080/00952990.2021.1969659. Epub 2021 Nov 9. PMID 34752714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with opioid use disorder who were voluntarily seeking treatment were eligible to enroll.
Pre-assignment Details: Two subjects were randomized, but did not receive study drug. Four subjects attempted enrollment at multiple sites. The data collected on these subjects during their second enrollment was excluded from the efficacy analyses.
Period: Overall Study
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Started | 126 | 126 | 126
Completed | 27 | 23 | 18
Not Completed | 99 | 103 | 108
Not completed — Adverse Event | 1 | 3 | 2
Not completed — Lost to Follow-up | 40 | 51 | 55
Not completed — Noncompliance with study drug | 0 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Protocol Violation | 4 | 2 | 3
Not completed — Withdrawal by Subject | 37 | 27 | 29
Not completed — Lack of Efficacy | 14 | 16 | 15
Not completed — Duplicate Patient | 1 | 0 | 0
Not completed — Patient not Stable | 0 | 1 | 0
Not completed — Incarceration | 0 | 1 | 0
Not completed — Failed Naloxone Challenge | 0 | 1 | 0
Not completed — Transportation Issues | 0 | 0 | 1
Not completed — Subject did not want last Vivitrol Injec | 0 | 0 | 1
Not completed — Noncompliance with Protocol | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety population included all subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B | Total
Number analyzed (Participants) | 126 | 126 | 126 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (10.68) | 37.5 (9.21) | 36.5 (10.38) | 38.0 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 47 | 42 | 129
  Male | 86 | 79 | 84 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 11 | 16 | 47
  Not Hispanic or Latino | 106 | 115 | 110 | 331
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 25 | 24 | 76
  White | 95 | 91 | 93 | 279
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 126 | 378

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Receive and Tolerate a VIVITROL Injection
Description: Toleration to the injection was demonstrated by mild opioid withdrawal symptoms (Clinical Opiate Withdrawal Scale [COWS] </=12 or Subjective Opiate Withdrawal Scale [SOWS] </=10) following VIVITROL administration. The COWS is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal. The SOWS is a 16-item self-report questionnaire designed to measure the severity of opioid withdrawal symptoms. The subject rates the intensity of symptoms using a 5-point scale. The range of SOWS scores is 1-10 (mild); 11-20 (moderate); and 21-30 (severe).
Time Frame: 1 week
Population: The Full Analysis Set (FAS) includes all subjects in the Safety Population (randomized subjects who received at least 1 dose of study drug), excluding the second enrollment of duplicate subjects (those subjects who enrolled multiple times in the same study).
Measure: Count of Participants; unit: Participants
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 124 | 126 | 124
Participants | 57 | 51 | 57
Statistical Analysis 1: Comparison: NTX/BUP vs PBO-N/PBO-B; Test type: Superiority; p = 0.940, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.61 to 1.70], Standard Error of Mean 0.264
Statistical Analysis 2: Comparison: NTX/PBO-B vs PBO-N/PBO-B; Test type: Superiority; p = 0.383, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.48 to 1.33], Standard Error of Mean 0.207

2. Secondary Outcome: Proportion of Days With COWS Peak Score of Less Than or Equal to 12 During the Treatment Period Prior to the VIVITROL Injection
Description: The Clinical Opiate Withdrawal Scale (COWS) is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal.
Time Frame: 1 week
Population: The Full Analysis Set (FAS) included all subjects in the Safety Population (randomized subjects who received at least 1 dose of study drug), excluding the second enrollment of duplicate subjects (those subjects who enrolled multiple times in the same study).
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 124 | 126 | 124
Number of days | 5.0 (2.23) | 4.5 (2.50) | 5.4 (2.02)

3. Secondary Outcome: Mean Peak COWS Score During Treatment Period Prior to VIVITROL Injection
Description: as for outcome 2
Time Frame: 1 week
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 124 | 126 | 124
score on a scale | 7.39 (3.726) | 7.78 (3.981) | 6.11 (3.044)

4. Secondary Outcome: Area Under the Curve (AUC) COWS Score During the Treatment Period Prior to VIVITROL Injection
Description: The Clinical Opiate Withdrawal Scale (COWS) is a clinician-rated questionnaire designed to measure 11 common opioid withdrawal signs or symptoms. The summed score provides information about the level of physical dependence on opioids. The range of COWS scores is 0-4 (none to minimal); 5-12 (mild); 13-24 (moderate); 25-36 (moderately severe); and 37-48 (severe withdrawal. To determine the daily AUC COWS score, a curve was generated by plotting the COWS scores against the time the test was taken. The area under this curve was calculated using the linear trapezoidal rule. For the total AUC COWS score, the AUCs calculated for each day during the treatment period were added together. To normalize for time, the total AUC COWS score was then divided by the number of days with daily AUC COWS score during the treatment period. The AUC COWS has a different range than the standard scale as it measures not the score itself, but the area under the curve of the score plotted against time.
Time Frame: The COWS was administered 4-6 times per day during the Treatment Period (Days 1-7)
Population: All randomized subjects who received at least 1 dose of study drug and had 1 post-baseline COWS measurement.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 124 | 126 | 124
Score on a scale | 955.7 (535.38) | 1004.8 (524.01) | 800.6 (403.01)

5. Secondary Outcome: Mean Score for Desire of Opioids During Treatment Period Prior to VIVITROL Injection
Description: The Desire for Opioids Visual Analog Scale (VAS) uses a 100-mm, horizontal linear scale, with 0 anchored on the left representing "no desire for opioids" and 100 anchored on the right representing "strongest imaginable desire for opioids". Subjects placed a vertical line on the scale to indicate their desire for opioids at that particular time.
Time Frame: 1 week
Population: All randomized subjects who received at least 1 dose of study drug and provided at least 1 post-baseline measureable VAS assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 123 | 124 | 123
score on a scale | 48.1 (27.61) | 52.0 (27.29) | 45.8 (26.03)

6. Secondary Outcome: Incidence of Adverse Effects
Description: The number of subjects who experienced treatment-emergent Adverse Events.
Time Frame: Up to 92 days
Population: The Safety Analysis Set was used to analyze this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 126 | 126 | 126
Participants | 44 | 31 | 48

7. Secondary Outcome: Area Under the Curve SOWS Score During the Treatment Period Prior to the VIVITROL Injection
Description: The Subjective Opiate Withdrawal Scale (SOWS) is a 16-item self-report questionnaire designed to measure the severity of opioid withdrawal symptoms. The subject rates the intensity of symptoms using a 5-point scale. The range of SOWS scores is 1-10 (mild); 11-20 (moderate); and 21-30 (severe). To determine the daily AUC SOWS score, a curve was generated by plotting the SOWS scores against the time the test was taken. The area under this curve was calculated using the linear trapezoidal rule. For the total AUC SOWS score, the AUCs calculated for each day during the treatment period were added together. To normalize for time, the total AUC SOWS score was then divided by the number of days with daily AUC SOWS score during the treatment period. The AUC SOWS has a different range than the standard scale as it measures not the score itself, but the area under the curve of the score plotted against time.
Time Frame: The SOWS was administered 4-6 times per day during the Treatment Period
Population: All randomized subjects who received at least 1 dose of study drug and had at least 1 post-baseline SOWS measurement.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
Number analyzed (Participants) | 111 | 114 | 112
Score on a scale | 9038.5 (6800.60) | 10,262.5 (7294.10) | 9160.3 (6873.56)

ADVERSE EVENTS:
Time Frame: Up to 92 days
Arm/Group | NTX/BUP | NTX/PBO-B | PBO-N/PBO-B
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/126 | 0/126
Serious Adverse Events (participants affected / at risk) | 2/126 | 1/126 | 2/126
Other Adverse Events (participants affected / at risk) | 18/126 | 12/126 | 19/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTX/BUP (N=126) | NTX/PBO-B (N=126) | PBO-N/PBO-B (N=126)
Panic Attack (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Alcohol use (Social circumstances) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTX/BUP (N=126) | NTX/PBO-B (N=126) | PBO-N/PBO-B (N=126)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 6 (7) | 9 (11)
Nausea (Gastrointestinal disorders) | 7 (8) | 4 (4) | 4 (5)
Anxiety (Psychiatric disorders) | 6 (6) | 4 (4) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.